CLINICAL TRIAL: NCT00707135
Title: A Phase Ib Study of Rapamycin (Sirolimus) in Patients With Advanced Malignancies
Brief Title: Rapamycin in Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13142A
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Rapamycin given once weekly in escalating doses. Higher dose levels will be split with the half the dose given on day 1 and half the dose on day 2 (24 hours later).
  Other Names: Rapamune; sirolimus

SUMMARY:
The goal of this study is to determine the rapamycin dose equivalent to the recommended phase II/III dose of temsirolimus and determine the observed toxicities and anti-tumor response of rapamycin in patients with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients with hematologic malignancies (lymphoma and CLL only) are eligible to participate in the phase Ib portion of the trial only. Patients must have relapsed or refractory disease that is no longer amenable to standard available therapy.
* At least 4 weeks since prior chemotherapy or radiation therapy
* Age >18 years
* ECOG performance status less than or equal to 2
* Life expectancy of greater than 3 months.
* Normal organ and marrow function as defined below:

  * No transfusions of packed red blood cells with 1 week of starting treatment. An absolute level of hemoglobin does not constitute an eligibility criterion but patients should be transfused as clinically indicated.
  * Leukocytes ≥ 3,000/μL
  * WBC ≥ 1,500/μL for patients with hematologic malignancies
  * ANC ≥ 1,500/μL (≥1,000/μL for patients with hematologic malignancies)
  * Absolute lymphocyte count ≥ 1000/µL
  * CD4 count ≥ 500/μL
  * Platelets ≥ 100,000/μL (≥50,000/μL for patients with hematologic malignancies)
  * Total bilirubin within normal institutional limits
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 times institutional upper limit of normal
  * Serum triglycerides ≤ 500 mg/dl
  * Creatinine within normal institutional limits OR
  * Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Not recovered from adverse events due to agents administered more than 4 weeks earlier.
* May not be receiving any other investigational agents.
* Uncontrolled brain metastases or malignancy. Patients with brain metastases or a malignant primary brain tumor must have stable neurologic status following local therapy (surgery or radiation) for at least 8 weeks from definitive therapy, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients cannot be receiving enzyme inducing anti-convulsants.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rapamycin.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, history of interstitial lung disease (including pneumonitis, bronchiolitis obliterans with organizing pneumonia, or pulmonary fibrosis) or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with severe immunodeficient states (as judged by the treating physician.
* Pregnant women, breast-feeding must be stopped
* HIV-positive patients are excluded due to possible pharmacokinetic interactions with rapamycin.
* Concurrent use of ketoconazole, cyclosporine, tacrolimus, and rifampin with rapamycin is not permissible. Concurrent use of rapamycin with diltiazem is allowed but should be done with caution or avoided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Dose level equivalent to recommended phase 2/3 dose of temsirolimus | 6 weeks
observed toxicities | 6 weeks
anti-tumor effect | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States